CLINICAL TRIAL: NCT00425100
Title: A 12-Week, Multicenter, Open-Label, Single-Arm Study To Evaluate The Effects Of Fesoterodine On Treatment Satisfaction And Symptom Relief In Overactive Bladder Patients.
Brief Title: A Clinical Trial To Assess Fesoterodine On Treatment Satisfaction And Symptom Improvement In Overactive Bladder Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0221007
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Results first posted 2009-02-10 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label-fesoterodine (Experimental): Single treatment study arm.
  Interventions: Drug: fesoterodine fumarate

INTERVENTIONS:
Drug: fesoterodine fumarate — 12 weeks of study treatment: Subjects received fesoterodine tablets 4 mg once daily for 4 weeks; thereafter, daily dosage was maintained at 4 mg or increased to 8 mg based on subject's and physician's subjective assessment of efficacy and tolerability.

SUMMARY:
To evaluate the effect of fesoterodine on patient satisfaction and overactive bladder (OAB) symptom relief in OAB patients who were dissatisfied with their prior therapy with tolterodine.

ELIGIBILITY:
Inclusion Criteria:

* OAB patients who present with OAB symptoms(≥8 micturitions and ≥3 urgency episodes per 24 h documented in the baseline bladder diary)
* OAB patients dissatisfied with their prior therapy with tolterodine

Exclusion Criteria:

* Patients with any contraindication to fesoterodine usage, e.g., urinary retention, gastric retention, uncontrolled narrow-angle glaucoma, or known hypersensitivity to the drug or its ingredients.
* Patients with significant hepatic and renal disease or other significant unstable diseases.
* OAB symptoms caused by neurological conditions, known pathologies of urinary tract, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (23):
  - Pfizer Investigational Site, Homewood, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Orangevale, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Aurora, Illinois
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Woodlane, New Jersey
  - Pfizer Investigational Site, Kingston, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Belgium (5):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Jette
  - Pfizer Investigational Site, Turnhout
- Costa Rica (2):
  - Pfizer Investigational Site, Alajuela Centro, Alajuela Province
  - Pfizer Investigational Site, San José
- Czechia (3):
  - Pfizer Investigational Site, Brno-Bohunice
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Prague
- Germany (7):
  - Pfizer Investigational Site, Alzey
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Duisburg
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, Muelheim A.d. Ruhr
  - Pfizer Investigational Site, München
- Poland (2):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Mysłowice
- Slovakia (5):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Malacky
  - Pfizer Investigational Site, Piešťany
  - Pfizer Investigational Site, Prešov
  - Pfizer Investigational Site, Skalica
- South Korea (5):
  - Pfizer Investigational Site, Bucheon-si, Gyunggi-do
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Jeonnam
  - Pfizer Investigational Site, Seoul
- Ukraine (5):
  - Pfizer Investigational Site, Chernivtsi
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Odesa
  - Pfizer Investigational Site, Zaporizhzhia

REFERENCES:
- [Derived] Wyndaele JJ, Goldfischer ER, Morrow JD, Gong J, Tseng LJ, Guan Z, Choo MS. Effects of flexible-dose fesoterodine on overactive bladder symptoms and treatment satisfaction: an open-label study. Int J Clin Pract. 2009 Apr;63(4):560-7. doi: 10.1111/j.1742-1241.2009.02035.x. PMID 19348029
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221007&StudyName=A%20Clinical%20Trial%20To%20Assess%20Fesoterodine%20On%20Treatment%20Satisfaction%20And%20Symptom%20Improvement%20In%20Overactive%20Bladder%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 59 centers (Belgium 5 centers, Costa Rica 2, Czech Republic 4, Germany 7, Republic of Korea 6, Poland 2, Slovakia 5, Ukraine 5, United States 23). Two centers in the United States did not randomize subjects.
Pre-assignment Details: 595 subjects were screened. Responses to a 5-day bladder diary (during a 2-week screening period) identified subjects who met all other entry criteria for enrollment for study treatment.
Groups:
- Open Label-fesoterodine: All enrolled subjects were treated with fesoterodine 4 mg once daily (QD) for 4 weeks followed by either 4 mg QD or 8 mg QD for the remaining 8 weeks of the study.
Period: Overall Study
Arm/Group | Open Label-fesoterodine
Started | 516
Completed | 463
Not Completed | 53
Not completed — Adverse Event | 36
Not completed — Lack of Efficacy | 4
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Open Label-fesoterodine
Number analyzed (Participants) | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 398
  Male | 118

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Micturition Episodes Per 24 Hours
Description: The mean number of micturitions per 24 hours is calculated as the total number of micturitions divided by the total number of diary days collected at that visit.
Time Frame: Baseline and Week 12
Population: Subjects in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 12 (last observation carried forward (LOCF)). The FAS included all subjects who took at least 1 dose of assigned study drug and contributed data to at least 1 baseline or post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 514 | 514
number of episodes | 12.7 (3.9) | 9.7 (3.4)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; Open-label study with statistical comparison between baseline and Week 12. Null hypothesis: The mean change from baseline in number of micturition episodes per 24 hours at Week 12 is equal to 0. The sample size was based on a statistical power for each of the three individual diary endpoints of .95 which would yield an overall power of 85%; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — All paired t-tests were performed with a two-sided test at significance level of 5%. Efficacy was claimed only when all 3 primary diary endpoints demonstrated statistical significance in change from baseline to Week 12; paired t-test comparing baseline with post-baseline values; Mean Difference (Net) = -3.0, 95% CI [-3.2 to -2.7], Standard Deviation 3.1

2. Primary Outcome: Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours
Description: The mean number of UUI episodes per 24 hours is calculated as the total number of micturitions with Bladder Sensation Scale (BSS) = 5 divided by the total number of diary days collected at that visit. BSS: 5 point scale measuring need to urinate from 1=no urgency to 5=unable to hold; leak urine.
Time Frame: Baseline and Week 12
Population: Subjects in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 12 (last observation carried forward (LOCF)). The FAS included all subjects who took at least 1 dose of assigned study drug and contributed data to at least 1 baseline or post-baseline efficacy assessment. Restricted to subjects with UUI at baseline >0.
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 256 | 256
number of episodes | 2.3 (2.8) | 0.6 (1.3)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; Open-label study with statistical comparison between baseline and Week 12. Null hypothesis: The mean change from baseline in number of urgency urinary incontinence per 24 hours is equal to 0. The sample size was based on a statistical power for each of the three individual diary endpoints of .95 which would yield an overall power of 85%; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 1, analysis 1]; paired t-test comparing baseline with post-baseline values; Mean Difference (Net) = -1.7, 95% CI [-2.0 to -1.4], Standard Deviation 2.4

3. Primary Outcome: Mean Number of Urgency Episodes Per 24 Hours
Description: The mean number of urgency episodes per 24 hours is calculated as the total number of micturitions with Bladder Sensation Scale (BSS) >= 3 divided by the total number of diary days collected at that visit. BSS: 5 point scale measuring need to urinate from 1=no urgency to 5=unable to hold; leak urine.
Time Frame: Baseline and Week 12
Population: Subjects in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 12 (last observation carried forward (LOCF)).The FAS included all subjects who took at least 1 dose of assigned study drug and contributed data to at least 1 baseline or post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 514 | 514
number of episodes | 10.0 (4.5) | 5.0 (4.7)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; Open-label study with statistical comparison between baseline and Week 12. Null hypothesis: The mean change from baseline in number of urgency episodes per 24 hours is equal to 0. The sample size was based on a statistical power for each of the three individual diary endpoints of .95 which would yield an overall power of 85%; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 1, analysis 1]; paired t-test comparing baseline with post-baseline values; Mean Difference (Net) = -5.0, 95% CI [-5.4 to -4.5], Standard Deviation 4.8

4. Primary Outcome: Number of Participants Reporting Satisfaction With Current Overactive Bladder (OAB) Treatment
Description: Number of Participants who responded satisfied = (very satisfied or somewhat satisfied) and dissatisfied = (somewhat dissatisfied or very dissatisfied) to the treatment satisfaction question.
Time Frame: Week 12
Population: Subjects in the Full Analysis Set (FAS) with non-missing value at Week 12. The FAS included all subjects who took at least 1 dose of assigned study drug and contributed data to at least 1 baseline or post-baseline efficacy assessment.
Measure: Number; unit: participants
Arm/Group | Open Label Week 12
Number analyzed (Participants) | 474
participants
  Satisfied (very satisfied or somewhat satisfied) | 378
  Neither dissatisfied nor satisfied | 42
  Dissatisfied (somewhat or very dissatisfied) | 54

5. Secondary Outcome: Nocturnal Micturitions Per 24 Hours
Description: Nocturnal micturitions (synonymous with the term "nighttime micturitions") were those recorded in the bedtime section of the bladder diary.
Time Frame: Baseline and Week 12
Population: Subjects in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 12 (LOCF). The FAS included all subjects who took at least 1 dose of assigned study drug and contributed data to at least 1 baseline or post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: number of nocturnal micturitions
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 514 | 514
number of nocturnal micturitions | 2.6 (1.6) | 1.8 (1.4)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2 sided paired t-test — P-value was not adjusted for multiple comparisons. All paired t-tests were performed with a two-sided test at significance level of 5%; Mean Difference (Net) = -0.8, Standard Deviation 1.2

6. Secondary Outcome: Severe Urgency Episodes Per 24 Hours
Description: Severe urgency episodes defined as Urinary Sensation Scale (USS) rating ≥4. Subjects rated the feeling of urgency associated with each micturition episode using USS provided in the bladder diary. Scale ranges from 1=no feeling of urgency to 5=unable to hold; leak urine; decrease indicates an improvement with respect to urgency symptoms.
Time Frame: Baseline and Week 12
Population: Subjects in the Full Analysis Set (FAS) with baseline severe urgency episodes >0 and non-missing numerical change from baseline to Week 12 (LOCF). The FAS included all subjects who took at least 1 dose of assigned study drug and contributed data to at least 1 baseline or post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 442 | 442
number of episodes | 5.0 (4.4) | 1.5 (2.7)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = -3.5, Standard Deviation 4.1

7. Secondary Outcome: Mean Rating on the Urinary Sensation Scale
Description: The mean rating was calculated as the sum of rating scores on the Urinary Sensation Scale divided by the total number of micturitions with non-missing rating at that visit. The scale ranges from 1 "no feeling of urgency" to 5 "unable to hold; leak urine."
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 514 | 514
scores on a scale | 3.2 (0.6) | 2.5 (0.7)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = -0.7, Standard Deviation 0.7

8. Secondary Outcome: Patient Perception of Bladder Condition (PPBC) Score
Description: The PPBC score ranges from 1 "no problems at all" to 6 "many severe problems."
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 487 | 487
scores on a scale | 4.9 (0.7) | 3.1 (1.2)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = -1.8, Standard Deviation 1.3

9. Secondary Outcome: Patient Perception of Bladder Condition (PPBC) Score at Week 12 Relative to Baseline (Categorical Change)
Description: Improvement: negative score change; No change: score change=0; Deterioration: positive score change
Time Frame: Baseline and Week 12
Population: Subjects in the Full Analysis Set (FAS) with non-missing change from baseline to Week 12 (LOCF). The FAS included all subjects who took at least 1 dose of assigned study drug and contributed data to at least 1 baseline or post-baseline efficacy assessment.
Measure: Number; unit: participants
Arm/Group | Open Label Week 12
Number analyzed (Participants) | 487
participants
  Improvement | 405
  No change | 72
  Deterioration | 10

10. Secondary Outcome: Urgency Perception Scale (UPS)
Description: UPS scores range from 0 ("I am usually not able to hold urine") to 2 ("I am usually able to finish what I am doing before going to the toilet [without leaking]").
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 485 | 485
scores on a scale | 0.8 (0.5) | 1.4 (0.6)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 0.5, Standard Deviation 0.7

11. Secondary Outcome: Urgency Perception Scale (UPS) at Week 12 Relative to Baseline (Categorical Change)
Description: Improvement: positive score change; No improvement: zero or negative score change
Time Frame: Baseline and Week 12
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Open Label Week 12
Number analyzed (Participants) | 485
participants
  Improvement | 237
  No improvement | 248

12. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) - Health Related Quality of Life (HRQL) Concern Domain
Description: Each item rated by subject on a Likert scale 1 (most favorable) to 6 (least favorable). Raw scores were transformed to a score from 0 to 100. Once transformed, higher scores represent more favorable outcome.
Time Frame: Baseline and Week 12
Population: Subjects in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 12. The FAS included all subjects who took at least 1 dose of assigned study drug and contributed data to at least 1 baseline or post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 470 | 470
scores on a scale | 50.5 (25.3) | 79.1 (21.2)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 28.6, Standard Deviation 26.4

13. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) - Health Related Quality of Life (HRQL) Coping Domain
Description: as for outcome 12
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 470 | 470
scores on a scale | 44.7 (25.3) | 75.3 (24.3)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 30.6, Standard Deviation 26.6

14. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) - Health Related Quality of Life (HRQL) Sleep Domain
Description: as for outcome 12
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 470 | 470
scores on a scale | 47.4 (25.5) | 72.3 (23.3)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 24.9, Standard Deviation 27.3

15. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) - Health Related Quality of Life (HRQL) Social Interaction Domain
Description: as for outcome 12
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 470 | 470
scores on a scale | 71.3 (23.5) | 88.1 (18.6)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 16.8, Standard Deviation 21.1

16. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) - Total Health Related Quality of Life (HRQL) Scale
Description: as for outcome 12
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 470 | 470
scores on a scale | 52.2 (21.8) | 78.3 (20.2)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 26.1, Standard Deviation 22.8

17. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) - Symptom Bother Scale
Description: Each item rated by subject on a Likert scale 1 (least symptom bother) to 6 (most symptom bother). Raw scores were transformed to a score from 0 to 100. Once transformed, higher scores represent less favorable outcome.
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 470 | 470
scores on a scale | 57.4 (18.7) | 28.6 (20.2)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = -28.7, Standard Deviation 22.7

18. Secondary Outcome: "Satisfaction With OAB Control" Module of Overactive Bladder (OAB) Treatment Satisfaction Questionnaire (TSQ) (OAB-S)
Description: Module coded on scale (1-very satisfied to 5-very dissatisfied). Coding reversed algorithmically & results transformed: total score range 0-100. Higher final response value associated with better satisfaction. Satisfied on TSQ = very or somewhat satisfied; Not satisfied on TSQ =very or somewhat dissatisfied or neither dissatisfied nor satisfied.
Time Frame: Week 12
Population: Population included subjects in FAS (described above) with non-missing values on OAB-S at Week 12, referred to in table below as All Subjects. Summary was presented for All Subjects and 2 subgroups, based on categorization for treatment satisfaction question used in primary endpoint assessing satisfaction.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Week 12
Number analyzed (Participants) | 473
scores on a scale
  All Subjects (N=473) | 74.7 (22.3)
  Subjects satisfied on TSQ (n=377) | 82.7 (14.0)
  Subjects not satisfied on TSQ (n=96) | 43.6 (21.5)

19. Secondary Outcome: Sum Rating on the Urinary Sensation Scale
Description: The sum rating per 24 hours was calculated as the mean rating score on the Urinary Sensation Scale multiplied by the mean number of micturitions per 24 hours at that visit. The scale ranges from 1 "no feeling of urgency" to 5 "unable to hold; leak urine."
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open Label Baseline | Open Label Week 12
Number analyzed (Participants) | 514 | 514
scores on a scale | 40.4 (15.6) | 25.2 (13.2)
Statistical Analysis 1: Comparison: Open Label Baseline vs Open Label Week 12; This is an open-label study with statistical comparison between baseline and Week 12; Test type: Superiority or Other; p < 0.0001, 2-sided paired t-test — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = -15.2, Standard Deviation 14.2

20. Secondary Outcome: Treated Subjects Reporting Satisfaction With Their Current OAB Treatment (Supportive Analysis)
Description: Number of participants who responded satisfied = (very satisfied or somewhat satisfied) or dissatisfied = (somewhat dissatisfied or very dissatisfied) to the treatment satisfaction question at Week 12 in the safety set.
Time Frame: Week 12
Population: Subjects in safety set included subjects who took at least one dose of study drug. Missing responses to the Treatment Satisfaction Question at Week 12 were imputed as not satisfied for calculating the most conservative treatment satisfaction.
Measure: Number; unit: participants
Arm/Group | Open Label Week 12
Number analyzed (Participants) | 516
participants
  Satisfied (very satisfied or somewhat satisfied) | 378
  Neither Dissatisfied nor Satisfied | 42
  Dissatisfied (somewhat or very dissatisfied) | 54
  Missing Response (imputed as dissatisfied) | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.